CLINICAL TRIAL: NCT06752941
Title: LOW-PV Continuation
Acronym: CONT-LOW-PV
Status: Recruiting | Type: Observational
Sponsor: FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS (Other)
Responsible Party: Sponsor
Other Study IDs: LOW-PV Continuation
Record Dates: First submitted 2024-12-17; First posted 2024-12-31 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Polycythemia Vera
Keywords: Ropeginterferon alfa-2b
MeSH Terms: conditions — Polycythemia Vera

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This multicenter longitudinal observational study focuses on Italian patients with Polycythemia Vera (PV) who were enrolled in the Low-PV RCT and continued receiving Ropeginterferon alfa-2b until the study's conclusion on March 31, 2023. It includes patients who were responders to Ropeginterferon alfa-2b after two years in the phase II randomized trial "LOW-PV." Data will be collected retrospectively every 6 months from March 31, 2023 to November 30, 2024 and prospectively from December 1, 2024 to March 31, 2026.

DETAILED DESCRIPTION:
Multicentre longitudinal observational Italian study of patients with Polycythemia Vera (PV) enrolled in Low-PV RCT and still receiving the experimental drug (i.e., Ropeginterferon alfa-2b) at study end (31-03-2023). Thirty-six patients who completed the Low-PV RCT and were responders to Interferon, continued treatment with the drug and are followed at their respective centers in Italy. The "LOW-PV Continuation" study aims to collect after 1,2,3 years the data on these patients, regardless of the treatment they were undergoing at the time of enrollment in the current study, after their informed consent. In details, data will be collected retrospectively from March 31, 2023 to November 2024 and prospectively from December 1, 2024 to March 31, 2026.

Given the descriptive nature of the study, no formal statistical hypothesis will be made.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the LOW-PV RCT study who continued to receive Ropeginterferon alfa-2b until the conclusion of the study on March 31, 2023. These patients will be included regardless of the treatment they are undergoing at the time of enrollment in the current study.
* Patients who have signed the written informed consent for study participation.

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty-six patients completed the Low-PV RCT and were still under treatment with Ropeg at study end. The "LOW-PV Continuation" study aim to update data of all these patients, regardless of the treatment they are undergoing at the time of enrollment in the current study, after having obtained their informed consent to participation.
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Maintenance of Treatment response | From date of randomization until the date of follow up assessed up to 6 months.
  Median HCT lower than 45% without disease progression

SECONDARY OUTCOMES:
Complete hematological (CHR) and clinical remission (CR) | From date of randomization until the date of follow up assessed up to 6 months
  Rate of Efficacy
Change in JAK2 variant allele frequency (VAF) since treatment start | From date of randomization until the date of follow up assessed up to 6 months
  Rate of Efficacy
Frequency of phlebotomies | From date of randomization until the date of follow up assessed up to 6 months
  Rate of Efficacy
Change in spleen size since treatment start | From date of randomization until the date of follow up assessed up to 6 months
  Rate of Efficacy
Incidence of any of the following: o arterial and venous thrombotic events; o hemorrhagic events; o disease related symptoms; o disease evolutions into myelofibrosis and acute leukemia; o secondary malignancies o death | During the follow up every 6months per patient.
  Rate of Efficacy
Discontinuation of Ropeginterferon alfa-2b for any reason | From date of randomization until the date of follow up assessed up to 6 months
  Rate of Efficacy
Incidence and grading of any adverse event related to Ropeginterferon alfa-2b | From date of randomization until the date of follow up assessed up to 6 months
  Rate of Safety

CONTACTS AND LOCATIONS:
Overall Officials: TIZIANO BARBUI, MD, Study Director — FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS
Locations (13):
- Italy (13):
  - Fondazione IRCCS Policlinico San Matteo, Divisione Ematologia, Pavia, Lombardy
  - Ospedale Borgo Roma, Divisione Ematologia, Verona, Veneto
  - ASST Papa Giovanni XXIII, SC Ematologia, Bergamo
  - Policlinico S. Orsola - Malpighi, UO Ematologia, Bologna
  - Azienda Ospedaliero Universitaria Careggi, SOD Ematologia, Florence
  - Fondazione IRCCS Cà Granda - Ospedale Maggiore Policlinico, SC Ematologia, Milan
  - Ospedale San Raffaele, Unità Operativa di Ematologia e Trapianto Midollo Osseo, Milan
  - Azienda Ospedaliera Universitaria Federico II di Napoli Divisione di Ematologia e Trapianti del Midollo, Napoli
  - Azienda Ospedaliero Universitaria Maggiore della Carità di Novara SCDU Ematologia, Novara
  - Policlinico Universitario Fondazione Agostino Gemelli, Roma
  - A.O.U. Città della Salute e della Scienza di Torino - Ospedale Molinette- S.C. Ematologia U, Torino
  - ASST Sette Laghi, Ospedale di Circolo e F. Macchi, Divisione UO Ematologia, Varese
  - Azienda ULSS 8 Berica - Ospedale San Bortolo, Divisione di Ematologia, Vicenza

IPD SHARING:
Plan to Share IPD: No